CLINICAL TRIAL: NCT06793514
Title: Efficacy and Safety of Oral Probiotics on Ocular Symptoms and Gut Microbiome of Children with Vernal Keratoconjunctivitis: a Double-blind Clinical Trial Study
Brief Title: Efficacy and Safety of Oral Probiotics on Ocular Symptoms and Gut Microbiome of Children with Vernal Keratoconjunctivitis
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Mohsen Pourazizi (Other)
Responsible Party: Sponsor-Investigator, Mohsen Pourazizi, Assistant Professor of Ophthalmology, Isfahan University of Medical Sciences
Organization: Isfahan University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IR.ARI.MUI.REC.1403.220
Record Dates: First submitted 2025-01-21; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Probiotic; Ocular Surface Disease; Ocular Diseases; Ocular Dryness; Gut Microbiome Dysbiosis; Gut -microbiota
Keywords: Probiotic; Vernal keratoconjunctivitis; Clinical trial; gut microbiome
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Case group: treatment with oral probiotics (Experimental): In the case group, the patients with vernal keratoconjunctivitis will receive oral probiotics within one month and outcomes will be assessed one month after probiotic therapy.
  Interventions: Drug: Probiotic
- Placebo group: treatment with placebo. (Placebo Comparator): In the placebo group, the patients with vernal keratoconjunctivitis will receive the placebo substance within one month and outcomes will be assessed one month after treatment.
  Interventions: Drug: Placebo Drug

INTERVENTIONS:
Drug: Probiotic — The experimental group will receive the oral probiotics (Lactobacillus casei, Lactobacillus rhamnosus, Lactobacillus acidophilus, Lactobacillus bulgaricus, Bifidobacterium breve, Bifidobacterium infantis, Streptococcus thermophiles) alongside with fructooligosaccharide (FOS), which is prepared in the concentration of 109 cfu by Bisot Khimr and is in the form of an edible sachet that can be dissolved in cold water, which is consumed once a day for one month. Sachets should be stored at a temperature of 2 to 8 degrees Celsius (in the refrigerator), which increases the useful life of probiotic bacteria and makes them more effective.
  Arms: Case group: treatment with oral probiotics
Drug: Placebo Drug — The placebo is also prepared in the form of probiotic supplement in the form of sachets with similar packaging by the bio-fermenting pharmaceutical company.
  Arms: Placebo group: treatment with placebo.

SUMMARY:
The primary goal of this study is to determine the effects of oral probiotics on the severity of ocular symptoms and the alterations of the gut microbiome of children (4-18 years old) with vernal keratoconjunctivitis. The current study will also assess the safety of oral probiotics among children with vernal keratoconjunctivitis. The main questions it aims to answer: 1- Does treatment with oral probiotics improve the severity of ocular symptoms in children with vernal keratoconjunctivitis? 2- Does treatment with oral probiotics alter the gut microbiome of children with vernal keratoconjunctivitis? Researchers will compare the ocular symptoms and gut microbiome between two groups receiving oral probiotics and placebo among children with vernal keratoconjunctivitis.

Participants The participants will receive the oral probiotics and placebo ever day for one month.

Record their regimen and keep a diary of their symptoms.

ELIGIBILITY:
Inclusion Criteria:1- Patients whose diagnosis of vernal keratoconjunctivitis is confirmed based on clinical criteria. 2-Patients with an age range of 4 to 18 years. 3-Patients who have not received drug treatment for vernal keratoconjunctivitis disease recently.

-

Exclusion Criteria:1-Having other eye diseases (except refractive error) 2-Change in the diagnosis of the disease during the study 3-Antibiotics, anti-inflammatory drugs, immunosuppressive drugs 4-History of known gastrointestinal diseases (such as IBD, Celiac,...) 5- History of digestive problems in the last two weeks 6- Lack of consent to participate in the study 7- Having an eye infection in the last one month 8- People who were athletes or involved in intense physical activity 9- Smoking, alcohol and drugs. 10- Using drugs that affect appetite, bowel movements, and nutrient absorption 11- Using prebiotics, probiotics or synbiotics in the last 3 months 12- People who have been on a diet to lose or gain weight in the last 3 months 13- People who have undergone gastrointestinal surgery. 14- Changing the patient's diagnosis in the course of treatment 15- Failure to follow up the patient at the specified times for the visit and assessment of the patient's bed 16- Taking fat-reducing drugs 17-Oral hypoglycemic drugs, insulin, antihypertensive drugs-18- Diuretics, laxatives, antacids 19-Food supplements in the last 3 months.

-

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
The severity of ocular symptoms | One month
  Clinical symptoms (itching, photosensitivity, burning and tearing) and signs (conjunctival hyperemia, chemosis, secretions, Trantas dots and superficial punctate keratitis) are evaluated using slit lamp examination and fluorescent staining and are scored from 0 to 3 points. (0=absence, 1=mild, 2=moderate, 3=severe). At the beginning of the study and one month after the start of the study, the total score of symptoms (range: 0-24) and the score of symptoms (range: 0-30) are calculated as the sum of the scores of each symptom.
Alterations of gut microbiota | One month
  The evaluation of gut microbiota will be conducted at baseline and one month after treatment using real time PCR.

SECONDARY OUTCOMES:
The recurrent rate of disease | Three month
  The recurrent rate of vernal keratoconjunctivitis will be determined after three months of treatment based on clinical manifestations.
The complications of treatment | Three month
  The potential complications (e.g., abdominal pain, vomiting, diarrhea, allergic reactions, etc) will be assessed one and three months after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Mohsen Pourazizi, Study Director — Isfahan University of Medical Sciences, Feiz Hospital, Isfahan Isfahan, Isfahan, Iran